CLINICAL TRIAL: NCT01661231
Title: BIOTRONIK - The Treatment of Iliac and Femoral Atherosclerotic Lesions Using the Self-expanding Astron and Pulsar-18 Stents (BIOFLEX-I Europe)
Brief Title: Study to Determine the Performance of the Astron and Pulsar-18 Stents in Europe
Acronym: BIOFLEX-I EU
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Active, not recruiting
Sponsor: Biotronik AG (Industry)
Collaborators: Biotronik, Inc. (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: C1106
Record Dates: First submitted 2012-08-02; First posted 2012-08-09 (Estimated); Last update posted 2017-02-03 (Estimated); Status verified 2017-02

CONDITIONS: Peripheral Artery Disease; Peripheral Vascular Disease
Keywords: Vascular intervention; Endovascular; Peripheral stent
MeSH Terms: conditions — Peripheral Arterial Disease; Peripheral Vascular Diseases

ARMS (1):
- Investigational Stents (Experimental): Device: Astron/Pulsar-18 Stents Implantation of self-expanding, bare-metal, nitinol stents for treatment of peripheral artery disease.
  Interventions: Device: Astron/Pulsar-18 stent

INTERVENTIONS:
Device: Astron/Pulsar-18 stent — Peripheral Vascular Intervention

SUMMARY:
BIOFLEX-I EU is the European arm of the BIOFLEX-I IDE study (NCT01319812). Data from BIOFLEX-I EU will be pooled with data in the IDE. The objective of this study is to separately demonstrate the clinical performance of BIOTRONIK's Astron and Pulsar-18 stents in the European arm of the BIOFLEX-I IDE (NCT01319812). The Pulsar-18 stent will be used for the treatment of femoro-popliteal lesions, located in the native superficial femoral artery (SFA) or proximal popliteal artery (PPA), while the Astron stent will be used for the treatment of the common or external iliac artery lesions.

ELIGIBILITY:
Inclusion Criteria:

* Age ≥ 18 years
* Willingness to comply with study follow-up requirements.
* Candidate for percutaneous transluminal angioplasty (PTA).
* Life-style limiting claudication or rest pain with an ABI ≤ 0.9 (resting or exercise). Thigh or toe brachial index (TBI) may be used / performed if ABI is inadequate.
* Written informed consent.
* One de novo, restenotic or occluded lesion representing a femoro-popliteal or iliac indication OR Two de novo, restenotic or occluded lesions representing one femoro-popliteal indication and one iliac indication on contralateral limbs - (i.e. one target lesion per limb).
* Lesions may be one solid lesion or a series of multiple, smaller lesions to be treated as one lesion.
* Subjects with bilateral, SFA/PPA disease (i.e. one SFA/PPA lesion per limb) are eligible for enrolment into the study. The target lesion will be selected at the investigator's discretion based on study eligibility criteria. The contralateral SFA/PPA intervention may be performed at the time of the index procedure (prior to treatment of study lesion); however, the use of an investigational treatment is prohibited. If the contralateral SFA/PPA intervention is not performed at the time of the index procedure, the intervention must be performed at least 30 days after the index procedure. The use of an investigational treatment for the contralateral intervention is prohibited.
* Subjects with bilateral, iliac disease (i.e. one iliac lesion per limb) are eligible for enrollment into the study. The target lesion will be selected at the investigator's discretion based on study eligibility criteria. The contralateral iliac intervention may be performed at the time of the index procedure; however, the use of an investigational treatment is prohibited. If the contralateral iliac intervention is not performed at the time of the index procedure, the intervention must be performed at least 30 days after the index procedure. The use of an investigational treatment for the subsequent contralateral intervention is also prohibited.
* Femoro-popliteal lesions must be located at least 1 cm distal to the profunda femoris artery and at least 3 cm above the knee joint (radiographic joint space).
* Iliac lesions must be located only in either the common or external iliac artery.
* Lesions must be treatable with a maximum of two stents.
* Angiographic evidence of ≥ 70% stenosis or occlusion (operator visual assessment).
* Lesion length ≤ 190 mm (if de novo or restenotic) or ≤ 100 mm (if occluded).
* Target vessel reference diameter: 2.5 to 6 mm (SFA/PPA) or 6 to 9 mm (iliac arteries) by visual estimate.
* Angiographic evidence of patent SFA and PPA (iliac indication) and angiographic evidence of at least one distal vessel runoff to the foot (both femoro-popliteal and iliac indications). Patent is defined as < 50% stenosis.
* For SFA/PPA intervention, a significant stenosis (> 70%) or occlusion of an ipsilateral, inflow artery (e.g. aortoiliac, common femoral) must be successfully treated with PTA and/or commercially-available stent just prior to treatment of the target lesion. Successful treatment is defined as no complications and less than 30% residual stenosis following intervention.

Exclusion Criteria:

* Subjects pregnant or planning to become pregnant during the course of the study.
* Life expectancy of less than one year.
* Rutherford-Becker category 5 or 6. Subjects with ulcers caused by venous disease may be enrolled in the study.
* Previously stented lesion(s) in the target vessel.
* Target lesion(s) received previous treatment within 30 days prior to enrollment.
* Prior peripheral vascular bypass surgery involving the target limb(s).
* Thrombophlebitis or deep vein thrombosis within the past 30 days.
* Known allergy to nitinol (nickel and/or titanium).
* Participation in any other clinical investigational device or drug study. Subjects may be concurrently enrolled in a post-market study, as long as the post-market study device, drug or protocol does not interfere with the investigational treatment or protocol of this study.
* Previous stroke or transient ischemic attack within the last three months prior to enrollment.
* Previous coronary or peripheral bypass surgery (non-target limb) within 30 days prior to enrollment.
* Intolerance to contrast agents that cannot be medically managed and/or intolerance to anti-platelet, anti-coagulant or thrombolytic medications.
* Refuses blood transfusions.
* Any medical condition, that in the opinion of the investigator, poses an unacceptable risk for implant of a stent according to the study indications.
* International Normalized Ratio (INR) ≥ 1.6
* Concomitant renal failure with serum creatinine level > 2.5 mg/dL
* Unresolved neutropenia (white blood cell count < 3,000 / µL) or thrombocytopenia (platelet count < 80,000 / µL) at the time of the index procedure.
* Unresolved bleeding disorder (INR ≥ 1.6) at the time of the index procedure.
* Presence of other ipsilateral, arterial lesions distal to the target lesion requiring treatment within 30 days of the index procedure (either before or after) or at the time of index procedure.
* Additional percutaneous interventional procedures (cardiac and/or peripheral) planned within 30 days after the index procedure.
* Presence of a complication following pre-dilation of target lesion.
* Presence of a target vessel/lesion that is excessively tortuous or calcified or is adjacent to an acute thrombus that is unresponsive to anti-thrombotic therapies.
* Target lesion is located within an aneurysm or associated with an aneurysm in the vessel segment either proximal or distal to the target lesion.
* Target lesion requires the use of cutting balloons, atherectomy or ablative devices.
* Subjects with less than single vessel runoff to the foot.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 456 (Estimated)
Dates: Start 2012-10; Primary Completion 2015-09 (Actual); Study Completion 2018-10 (Estimated)

PRIMARY OUTCOMES:
Primary Endpoint for the Astron Stent | 12 months
  A composite of the rate of procedure- or stent-related major adverse events (MAEs) at 12 months post-index procedure. The MAE rate includes 30-day mortality, along with 12-month rates of target lesion revascularization (TLR) and index limb amputation.
Clinical Primary Endpoint for the Pulsar-18 Stent | 30 days
  Freedom from procedure- or stent-related MAEs at 30 days post-index procedure. The MAE rate includes mortality, TLR and index limb amputation.
Performance Primary Endpoint for the Pulsar-18 Stent | 12 months
  Primary patency rate (defined as freedom from more than 50% restenosis) at 12 months post-index procedure, as measured by duplex ultrasound.

SECONDARY OUTCOMES:
Secondary Endpoint for the Pulsar-18 Stent | 30 days
  Contribution of the individual rates of mortality, TLR and index limb amputation at 30 days post-index procedure to the primary clinical endpoint for the Pulsar-18 stent group
Secondary Endpoint for the Astron Stent | 12 months
  Contribution of the individual rates of 30-day mortality and 12-month TLR and index limb amputation rates to the primary endpoint for the Astron stent.
Secondary Endpoint for the Pulsar-18 Stent | 12 months
  Evaluate the MAE rate of the Pulsar-18 stent group at 12 months post-index procedure, along with the contribution the individual rates of 30-day mortality and 12-month TLR and index limb amputation rates to the overall MAE rate
Secondary Endpoint for the Pulsar-18 Stent | 12 months
  Evaluate the stent fracture rate for the Pulsar-18 stent group at 12 months post-index procedure.
Secondary Endpoint for the Astron Stent | 12 months
  Evaluate the primary patency rate for the Astron stent at 12 months post-index procedure.
Secondary Endpoint for Both the Astron and Pulsar-18 Stents | 12 months
  Evaluate the primary assisted patency rate for the Astron stent and the Pulsar-18 stent group at 12 months post-index procedure.
Secondary Endpoint for Both the Astron and Pulsar-18 Stents | 12 months
  Evaluate the secondary patency rate for the Astron stent and the Pulsar-18 stent group at 12 months post-index procedure.
Secondary Endpoint for Both the Astron and Pulsar-18 Stents | 30 days
  Evaluate the 30-day clinical success of the procedure.
Secondary Endpoint for Both the Astron and Pulsar-18 Stents | 12 months
  Compare the ABI measurement(s) of the treated limb(s) between baseline and 12 months post-index procedure.
Secondary Endpoint for Both the Astron and Pulsar-18 Stents | 12 months
  Compare the scores on the Walking Impairment Questionnaire between baseline and 12 months post-index procedure.
Secondary Endpoint for Both the Astron and Pulsar-18 Stents | 30 days
  Evaluate the acute procedural success of the Astron stent and the Pulsar-18 stent group
Secondary Endpoint for Both the Astron and Pulsar-18 stents | 12 months
  Evaluate the rates of all individual adverse event types that are not included in the primary endpoint analyses for the Astron and Pulsar-18 stents
Comparison of Endpoints Results Between Short and Long Lesions for Pulsar-18 Stent | 12 months
  Compare the primary and secondary endpoint results between evaluable subjects in the Pulsar-18 stents with lesions from 20 mm to 140 mm in length and evaluable subjects with lesions from 141 mm to 190 mm in length.
Comparison of Endpoints Results Between Occlusive and Non-occlusive Lesions for Astron and Pulsar-18 Stents | 12 months
  Compare the primary and secondary endpoint results between evaluable subjects treated for occlusive lesions (100% stenosis) and evaluable subjects treated for non-occlusive lesions (70% - 99% stenosis) for the Astron stent and the Pulsar-18 stent group.
Secondary Endpoint for Both the Astron and Pulsar-18 Stents | 12 months
  Compare the distance walked during the six-minute walk test between baseline and 12 months post-index procedure

CONTACTS AND LOCATIONS:
Overall Officials: Marianne Brodmann, MD, Principal Investigator — Medical University of Graz, Graz, Austria
Locations (7):
- Medical University of Graz, Graz, Austria
- Belgium (3):
  - Imelda Ziekenhuis, Bonheiden
  - AZ St.-Blasius Hospital, Dendermonde
  - Regionaal Ziekenhuis Heilig Hart Tienen, Tienen
- Germany (2):
  - Klinikum Arnsberg, Karolinen Hospital Huesten, Arnsberg
  - Universitätsklinikum Münster, Münster
- University Hospital of Bern, Bern, Switzerland

REFERENCES:
- See also: Investigational Device Exemption Study to Determine the Safety and Efficacy of the Astron and Pulsar Stents (BIOFLEX-I) — http://clinicaltrials.gov/ct2/show/NCT01319812